CLINICAL TRIAL: NCT02377622
Title: Comparison of the Clinical Performance of 2 THERANOVA 400 Dialyzer Prototypes in HD With a High-Flux Dialyzer in HD and a High-Flux Dialyzer in hvHDF - A Pilot Study
Brief Title: Clinical Performance Comparison of 2 THERANOVA 400 Dialyzer Prototypes in HD With High-Flux Dialyzers in HD and hv HDF Mode
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1407-001
Record Dates: First submitted 2015-02-03; First posted 2015-03-03 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- THERANOVA 400 dialyzer prototype AA (Experimental): THERANOVA 400 dialyzer prototype AA in hemodialysis
  Interventions: Device: THERANOVA 400 dialyzer prototype AA
- THERANOVA 400 dialyzer prototype BB (Experimental): THERANOVA 400 dialyzer prototype BB in hemodialysis
  Interventions: Device: THERANOVA 400 dialyzer prototype BB
- FX CorDiax 80 dialyzer (Active Comparator): FX CorDiax 80 dialyzer in hemodialysis
  Interventions: Device: FX CorDiax 80 Dialyzer
- FX CorDiax 800 dialyzer (Active Comparator): FX CorDiax 800 dialyzer in high volume hemodiafiltration
  Interventions: Device: FX CorDiax 800 Dialyzer

INTERVENTIONS:
Device: THERANOVA 400 dialyzer prototype AA
  Arms: THERANOVA 400 dialyzer prototype AA
Device: THERANOVA 400 dialyzer prototype BB
  Arms: THERANOVA 400 dialyzer prototype BB
Device: FX CorDiax 80 Dialyzer
  Arms: FX CorDiax 80 dialyzer
Device: FX CorDiax 800 Dialyzer
  Arms: FX CorDiax 800 dialyzer

SUMMARY:
The study investigates the performance of a new dialyzer (Theranova 400) containing a membrane with increased pore sizes. The performance will be determined by the removal of middle molecules (with different molecular size) from the blood compartment. Two different Theranova 400 prototypes (AA and BB) operated in hemodialysis mode will be compared with a Cordiax Fx-80 dialyzer, operated in hemodialysis mode, and with a Cordiax Fx-800, operated in high volume hemodiafiltration mode. Safety events and albumin loss into the dialysate will be monitored

ELIGIBILITY:
Inclusion Criteria:

1. Patient has end-stage renal disease (Chronic kidney disease stage 5D)
2. Patient is 18 years of age or older
3. Patient is male or female
4. Patient, if female, is non-pregnant; and if capable of becoming pregnant, will be using a medically acceptable means of contraception during participation in the study 5 .Patient has been receiving HD or HDF therapy for >3 months prior to study enrollment and is expected to survive for at least 12 months after enrollment.

6. Patient has a stable functioning native fistula 7. Patient is willing to comply with the study requirements for therapy during the entire study treatment period 8. Patient is capable fo providing written informed consent to participate in the study

Exclusion Criteria:

1. Patient is undergoing single-needle dialysis
2. Patient has an known abnormal k/λ ratio (less than 0.37, or greater than 3.1)
3. Patient has a known active infection and is currently receiving antibiotic treatment
4. Patient has known active cancer
5. Patient has a known positive serology test for human immunodeficiency virus (HIV) or hepatitis B,C or E
6. Patient has a known serious hemostasis disorder
7. Patient has a known monoclonal gammopathy
8. Patient has a known polyclonal gammopathy
9. Patient has a unstable condition as judged by the treating physician based on medical history, physical examination and laboratory testing including (but not limited to) any of the following:

   * Myocardial infarction within the last 3 months
   * Tachyarrhythmia or bradyarrhythmia absoluta
   * Unstable angina pectoris
   * Left ventricular ejection fraction <30%
   * Significant pericardial disease
10. Patient has any other known comorbidity that could, in the opinion of the Investigator, potentially conflict with the study purpose or procedure
11. Patient has a known significant psychiatric disorder or mental disability that could interfere with the patient's ability to provide informed consent and/or comply with protocol procedures
12. Patient has a history of non-compliance with the dialysis prescription, as assessed by the Investigator
13. Patient has participated in another interventional clinical study in the past 3 months, or is currently participating in another interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Overall clearance of lambda FLC clearance | Five (5) hours ( for each mid-week dialysis session)
  Blood and dialysate
Overall albumin loss | Five (5) hours (for each mid-week dialysis session)
  Dialysate

SECONDARY OUTCOMES:
Types and frequency of adverse events and device deficiencies as a measure of safety and dialyzer tolerability | Average 60 days (continuously, from signature of informed consent form until 1 week after last hemodialysis session with an experimental or active comparator product)
  All adverse events and device deficiencies will be recorded
Clearance of other middle sized molecules | Five (5) hours (for each mid-week dialysis session)
  Blood and dialysate
Hematology ( blood cell counts; hematocrit and hemoglobin) | Five (5) hours ( for each mid-week dialysis session)
  Blood

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Böhler, Manager, Study Director — Life Sciences & Operations, Gambro Dialysatoren GmbH (a subsidiary of Baxter International Inc.)
Locations (1):
- Dialysexentrum Elsenfeld, Elsenfeld, Germany

REFERENCES:
- [Result] Kirsch AH, Lyko R, Nilsson LG, Beck W, Amdahl M, Lechner P, Schneider A, Wanner C, Rosenkranz AR, Krieter DH. Performance of hemodialysis with novel medium cut-off dialyzers. Nephrol Dial Transplant. 2017 Jan 1;32(1):165-172. doi: 10.1093/ndt/gfw310. PMID 27587605
- [Result] Kirsch AH, Rosenkranz AR, Lyko R, Krieter DH. Effects of Hemodialysis Therapy Using Dialyzers with Medium Cut-Off Membranes on Middle Molecules. Contrib Nephrol. 2017;191:158-167. doi: 10.1159/000479264. Epub 2017 Sep 14. PMID 28910799